CLINICAL TRIAL: NCT05874089
Title: The Role of VSL#3® in the Treatment of Fatigue and Other Symptoms in Long Covid-19 Syndrome: a Randomized, Double-blind, Placebo-controlled Study (DELong#3)
Brief Title: VSL#3® vs Placebo in the Treatment of Fatigue and Other Symptoms in Long Covid (DELong#3)
Acronym: DELong#3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Flavio Caprioli, Associate Professor of Gastroenterology, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DELong#3
Record Dates: First submitted 2023-05-21; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Long COVID
Keywords: Long Covid; Fatigue; Gut Microbioma; Dysbiosis; COVID-19; Coronavirus Infections
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue; Dysbiosis; COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This is a single-center randomized, double-blind, placebo-controlled trial. Patients will be recruited from Long Covid out-patient Clinics at Policlinico di Milano Hospital (Milan, Italy) and randomly assigned (1:1) to receive VSL#3® or placebo at the dosage of 2 sachets/die for 28 days. Fasting blood samples and feces will be collected before (t0) and after treatment (t4). Primary and secondary outcome will be assessed at baseline (t0), end of treatment (t4) and end of follow-up (t8) using validated questionnaires (i.e. CFS- Chalder Fatigue Scale; HAD- Hospital Anxiety and Depression Scale, SF36 - Short Form Health Survey, Structured Assessment of Gastrointestinal Symptoms Scale - SAGIS; Symptoms Check List 12 - SCL-12; Karnofsky Performance Status - KPS; Visual Analogue Scale- VAS). Subject participation in this study will be approximately 10 weeks, which include 2-weeks screening/run in period, 4-weeks treatment period and 4-weeks follow-up period.
Who Masked: Participant, Investigator
Masking Description: Double blinding is achieved by packaging probiotics and placebo in the same sealed and consecutively numbered containers with sachets similar in packaging, smell, and taste. All study participants and on-site study personnel will remain masked for the treatment allocation (randomized controlled trial phase) until database lock and signature of the statistical analysis plan.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VSL#3® (Active Comparator): VSL#3® 450 billion sachets, two sachets per day (900 billion of bacteria per day) for 28 days
  Interventions: Dietary Supplement: VSL#3®
- Placebo (Placebo Comparator): Placebo sachets, two sachets per day for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3® — VSL#3® 450 billions/sachets
  Arms: VSL#3®
Dietary Supplement: Placebo — Placebo sachets with maltose, cornstarch and dioxide
  Other Names: Placebo (for VSL#3®)
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effectiveness of VSL#3® in reducing Fatigue and other symptoms in Long Covid Syndrome compared to placebo.

DETAILED DESCRIPTION:
Long Covid syndrome is a chronic condition characterized by persistent symptoms experienced by individuals who have recovered from acute coronavirus disease (COVID-19). Among the various symptoms reported, fatigue stands out as a particularly burdensome and pervasive issue, significantly impacting the quality of life and daily functioning of Long Covid patients. Recent studies report that gut microbiota is altered during acute illness and not restored even after several months from recovery. Based on this evidence, modulation of intestinal microbiota can be considered as a possible therapeutic approach for Long Covid Syndrome. On this basis, the aim of this study is to evaluate efficacy of VSL#3® compared to placebo in reducing Fatigue in Long Covid Symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age >18; <65 yo
* Previous diagnosis of SARS-CoV-2 infection, documented by nasopharyngeal or antigenic molecular swab;
* Not currently be in quarantine or isolation;
* No antibiotics treatment in the 30 days prior to the trial;
* Chalder Fatigue Scale (in dichotomous form)>=4 possibly associated with signs and symptoms of Long COVID-19 syndrome: signs and symptoms that develop during or after SARS-CoV-2 infection, which persist for more than 4 weeks and are not reasonably explained otherwise; signs and symptoms include: fatigue, sleep disturbances, cognitive deficits (i.e. brain fogging, loss of concentration and memory, anxiety, depression), strength deficits, arthralgias and myalgias, gastroenterological alterations (reduced appetite, nausea, changes in bowel habits, abdominal pain

Exclusion Criteria:

* Cardiovascular and pulmonary disease with moderately severe organ dysfunction (NYHA>2, Borg scale>=2);
* Decompensated endocrine and metabolic diseases (child cirrhosis >= B, decompensated hypo/hyperthyroidism, decompensated hypoadrenalism)
* Diagnosis of FM, CFS/ME, and/or IBS prior to SARS-CoV-2 infection;
* Confirmed diagnoses of neurological pathologies, psychiatric diseases and cognitive disorders prior to SARS-CoV-2 infection;
* Previous confirmed diagnosis of chronic musculoskeletal pathologies prior to prior to SARS-CoV-2 infection;
* Refusal to participate in the study / refusal to process personal data;
* Pregnancy or breastfeeding;
* Addiction to alcohol or drugs in previous years;
* Use of other probiotics during the trial;
* Use of antibiotics during the trial and in the previous 30 days;
* Substantial change of diet during the trial;
* Participation in another clinical study in the previous 30 days or previous participation in this same trial;
* Known intolerance/hypersensitivity to the investigational drug or to the excipients of the placebo formulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-09-03 (Estimated); Study Completion 2023-11-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of Fatigue variation after 4 weeks of treatment (t4) | 4 weeks
  To determine if there is a statistically significant variation in the scores on the Chalder Fatigue Scale between the treated group and the placebo group after 4 weeks of treatment (t4)

SECONDARY OUTCOMES:
Assessment of Fatigue variation after 4 weeks of follow-up (t8) | 8 weeks
  To determine if there is a statistically significant difference in the scores on the Chalder Fatigue Scale between the treated group and the placebo group after 4 weeks of follow-up
Evaluation of Anxiety and Depression variation after 4 weeks of treatment (t4) | 4 weeks
  To determine if there is a statistically significant difference in the scores on the Hospital Anxiety and Depression Scale (HAD) between the treated group and to the placebo group after 4 weeks of treatment
Evaluation of Anxiety and Depression variation after 4 weeks of follow-up (t8) | 8 weeks
  To determine if there is a statistically significant difference in the scores on the Hospital Anxiety and Depression Scale (HAD) between the treated group and to the placebo group after 4 weeks of follow-up
Measurement of Quality of Life variation after 4 weeks of treatment (t4) | 4 weeks
  To determine if there is a statistically significant difference in the scores on the Short Form Health Survey (SF)-36 between the treated group and placebo group after 4 weeks of treatment
Measurement of Quality of Life variation after 4 weeks of follow-up (t8) | 8 weeks
  To determine if there is a statistically significant difference in the scores on the Short Form Health Survey (SF)-36 between the treated group and the placebo group after 4 weeks of follow-up
Assessment of Gastrointestinal Symptoms variation after 4 weeks of treatment (t4) | 4 weeks
  To determine if there is a statistically significant difference in the scores on the Structured Assessment of Gastrointestinal Symptoms Scale (SAGIS) between the placebo group and the treated group after 4 weeks of treatment
Assessment of Gastrointestinal Symptoms variation after4 weeks of follow-up (t8) | 8 weeks
  To determine if there is a statistically significant difference in the scores on the Structured Assessment of Gastrointestinal Symptoms Scale (SAGIS) between the placebo group and the treated group after 4 weeks of follow-up
Analysis of Somatization variation after 4 weeks of treatment (t4) | 4 weeks
  To identify the level of somatization of symptoms by comparing the scores on the SCL-12 for the somatization of Symptom Checklist-90 (SCL-90) between the treated group and the placebo group after 4 weeks of treatment
Analysis of Somatization variation after 4 weeks of treatment (t4) | 8 weeks
  To identify the level of somatization of symptoms by comparing the scores on the SCL-12 for the somatization of Symptom Checklist-90 (SCL-90) between the treated groups and the placebo group after 4 weeks of follow-up
Evaluation of Functional Status variation after 4 weeks of treatment (t4) | 4 weeks
  To assess the general functional status of the patients by comparing the scores on the Karnofsky Performance Status (KPS) Scale between the treated group and the placebo group after 4 weeks of treatment
Evaluation of Functional Status variation after 4 weeks of follow-up (t8) | 8 weeks
  To assess the general functional status of the patients by comparing the scores on the Karnofsky Performance Status (KPS) Scale between the treated group and the placebo group after 4 weeks of follow-up
Physician's Assessment of General Health variation after 4 weeks of treatment (t4) | 4 weeks
  To determine the physician's evaluation of the patient's general state of health using a visual-analogue scale (VAS) and comparing it between the treated group and the placebo group after 4 weeks of treatment
Physician's Assessment of General Health variation after 4 weeks of follow-up (t8) | 8 weeks
  To determine the physician's evaluation of the patient's general state of health using a visual-analogue scale (VAS) and comparing it between the treated group and the placebo group after 4 weeks of follow-up
Analysis of PBMC and Serum Expression of inflammatory mediators at baseline (t0) and after 4 weeks of treatment (t4) | 4 weeks
  Evaluation of multiple cytokines and chemokines in plasma samples and of immune cell phenotypes in peripheral blood mononuclear cells (PBMCs)
Investigation of Faecal Microbiota Variation after 4 weeks of treatment (t4) | 4 weeks
  To analyze the variation of the bacterial component of the faecal microbiota in terms of alpha and beta diversity and explore its correlation with clinical response on fatigue in both the placebo group and the treated group by using. Shotgun metagenomics and 16S sequencing of faecal samples at baseline and after 4 weeks of treatment (t4) generate serial gut microbial taxonomic and bacterial functional profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Caprioli, MD, PhD, Study Director — Fondazione IRCCS Cà Granda, Ospedale Policlinico di Milano
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ancona G, Alagna L, Alteri C, Palomba E, Tonizzo A, Pastena A, Muscatello A, Gori A, Bandera A. Gut and airway microbiota dysbiosis and their role in COVID-19 and long-COVID. Front Immunol. 2023 Mar 8;14:1080043. doi: 10.3389/fimmu.2023.1080043. eCollection 2023. PMID 36969243
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Ceban F, Ling S, Lui LMW, Lee Y, Gill H, Teopiz KM, Rodrigues NB, Subramaniapillai M, Di Vincenzo JD, Cao B, Lin K, Mansur RB, Ho RC, Rosenblat JD, Miskowiak KW, Vinberg M, Maletic V, McIntyre RS. Fatigue and cognitive impairment in Post-COVID-19 Syndrome: A systematic review and meta-analysis. Brain Behav Immun. 2022 Mar;101:93-135. doi: 10.1016/j.bbi.2021.12.020. Epub 2021 Dec 29. PMID 34973396
- [Background] Chen Y, Gu S, Chen Y, Lu H, Shi D, Guo J, Wu WR, Yang Y, Li Y, Xu KJ, Ding C, Luo R, Huang C, Yu L, Xu M, Yi P, Liu J, Tao JJ, Zhang H, Lv L, Wang B, Sheng J, Li L. Six-month follow-up of gut microbiota richness in patients with COVID-19. Gut. 2022 Jan;71(1):222-225. doi: 10.1136/gutjnl-2021-324090. Epub 2021 Apr 8. No abstract available. PMID 33833065
- [Background] Choutka J, Jansari V, Hornig M, Iwasaki A. Unexplained post-acute infection syndromes. Nat Med. 2022 May;28(5):911-923. doi: 10.1038/s41591-022-01810-6. Epub 2022 May 18. PMID 35585196
- [Background] Davis HE, McCorkell L, Vogel JM, Topol EJ. Long COVID: major findings, mechanisms and recommendations. Nat Rev Microbiol. 2023 Mar;21(3):133-146. doi: 10.1038/s41579-022-00846-2. Epub 2023 Jan 13. PMID 36639608
- [Background] Farsi Y, Tahvildari A, Arbabi M, Vazife F, Sechi LA, Shahidi Bonjar AH, Jamshidi P, Nasiri MJ, Mirsaeidi M. Diagnostic, Prognostic, and Therapeutic Roles of Gut Microbiota in COVID-19: A Comprehensive Systematic Review. Front Cell Infect Microbiol. 2022 Mar 4;12:804644. doi: 10.3389/fcimb.2022.804644. eCollection 2022. PMID 35310853
- [Background] Fernandez-de-Las-Penas C, Rodriguez-Jimenez J, Cancela-Cilleruelo I, Guerrero-Peral A, Martin-Guerrero JD, Garcia-Azorin D, Cornejo-Mazzuchelli A, Hernandez-Barrera V, Pellicer-Valero OJ. Post-COVID-19 Symptoms 2 Years After SARS-CoV-2 Infection Among Hospitalized vs Nonhospitalized Patients. JAMA Netw Open. 2022 Nov 1;5(11):e2242106. doi: 10.1001/jamanetworkopen.2022.42106. PMID 36378309
- [Background] Giannos P, Prokopidis K. Gut dysbiosis and long COVID-19: Feeling gutted. J Med Virol. 2022 Jul;94(7):2917-2918. doi: 10.1002/jmv.27684. Epub 2022 Mar 7. No abstract available. PMID 35233795
- [Background] Global Burden of Disease Long COVID Collaborators; Wulf Hanson S, Abbafati C, Aerts JG, Al-Aly Z, Ashbaugh C, Ballouz T, Blyuss O, Bobkova P, Bonsel G, Borzakova S, Buonsenso D, Butnaru D, Carter A, Chu H, De Rose C, Diab MM, Ekbom E, El Tantawi M, Fomin V, Frithiof R, Gamirova A, Glybochko PV, Haagsma JA, Haghjooy Javanmard S, Hamilton EB, Harris G, Heijenbrok-Kal MH, Helbok R, Hellemons ME, Hillus D, Huijts SM, Hultstrom M, Jassat W, Kurth F, Larsson IM, Lipcsey M, Liu C, Loflin CD, Malinovschi A, Mao W, Mazankova L, McCulloch D, Menges D, Mohammadifard N, Munblit D, Nekliudov NA, Ogbuoji O, Osmanov IM, Penalvo JL, Petersen MS, Puhan MA, Rahman M, Rass V, Reinig N, Ribbers GM, Ricchiuto A, Rubertsson S, Samitova E, Sarrafzadegan N, Shikhaleva A, Simpson KE, Sinatti D, Soriano JB, Spiridonova E, Steinbeis F, Svistunov AA, Valentini P, van de Water BJ, van den Berg-Emons R, Wallin E, Witzenrath M, Wu Y, Xu H, Zoller T, Adolph C, Albright J, Amlag JO, Aravkin AY, Bang-Jensen BL, Bisignano C, Castellano R, Castro E, Chakrabarti S, Collins JK, Dai X, Daoud F, Dapper C, Deen A, Duncan BB, Erickson M, Ewald SB, Ferrari AJ, Flaxman AD, Fullman N, Gamkrelidze A, Giles JR, Guo G, Hay SI, He J, Helak M, Hulland EN, Kereselidze M, Krohn KJ, Lazzar-Atwood A, Lindstrom A, Lozano R, Malta DC, Mansson J, Mantilla Herrera AM, Mokdad AH, Monasta L, Nomura S, Pasovic M, Pigott DM, Reiner RC Jr, Reinke G, Ribeiro ALP, Santomauro DF, Sholokhov A, Spurlock EE, Walcott R, Walker A, Wiysonge CS, Zheng P, Bettger JP, Murray CJL, Vos T. Estimated Global Proportions of Individuals With Persistent Fatigue, Cognitive, and Respiratory Symptom Clusters Following Symptomatic COVID-19 in 2020 and 2021. JAMA. 2022 Oct 25;328(16):1604-1615. doi: 10.1001/jama.2022.18931. PMID 36215063
- [Background] Guo C, Che X, Briese T, Ranjan A, Allicock O, Yates RA, Cheng A, March D, Hornig M, Komaroff AL, Levine S, Bateman L, Vernon SD, Klimas NG, Montoya JG, Peterson DL, Lipkin WI, Williams BL. Deficient butyrate-producing capacity in the gut microbiome is associated with bacterial network disturbances and fatigue symptoms in ME/CFS. Cell Host Microbe. 2023 Feb 8;31(2):288-304.e8. doi: 10.1016/j.chom.2023.01.004. PMID 36758522
- [Background] Li N, Ma WT, Pang M, Fan QL, Hua JL. The Commensal Microbiota and Viral Infection: A Comprehensive Review. Front Immunol. 2019 Jul 4;10:1551. doi: 10.3389/fimmu.2019.01551. eCollection 2019. PMID 31333675
- [Background] Marasco G, Cremon C, Barbaro MR, Cacciari G, Falangone F, Kagramanova A, Bordin D, Drug V, Miftode E, Fusaroli P, Mohamed SY, Ricci C, Bellini M, Rahman MM, Melcarne L, Santos J, Lobo B, Bor S, Yapali S, Akyol D, Sapmaz FP, Urun YY, Eskazan T, Celebi A, Kacmaz H, Ebik B, Binicier HC, Bugdayci MS, Yagci MB, Pullukcu H, Kaya BY, Tureyen A, Hatemi I, Koc ES, Sirin G, Caliskan AR, Bengi G, Alis EE, Lukic S, Trajkovska M, Hod K, Dumitrascu D, Pietrangelo A, Corradini E, Simren M, Sjolund J, Tornkvist N, Ghoshal UC, Kolokolnikova O, Colecchia A, Serra J, Maconi G, De Giorgio R, Danese S, Portincasa P, Di Sabatino A, Maggio M, Philippou E, Lee YY, Salvi D, Venturi A, Borghi C, Zoli M, Gionchetti P, Viale P, Stanghellini V, Barbara G; GI-COVID19 study group. Post COVID-19 irritable bowel syndrome. Gut. 2022 Dec 9:gutjnl-2022-328483. doi: 10.1136/gutjnl-2022-328483. Online ahead of print. PMID 36591612
- [Background] Nagata N, Takeuchi T, Masuoka H, Aoki R, Ishikane M, Iwamoto N, Sugiyama M, Suda W, Nakanishi Y, Terada-Hirashima J, Kimura M, Nishijima T, Inooka H, Miyoshi-Akiyama T, Kojima Y, Shimokawa C, Hisaeda H, Zhang F, Yeoh YK, Ng SC, Uemura N, Itoi T, Mizokami M, Kawai T, Sugiyama H, Ohmagari N, Ohno H. Human Gut Microbiota and Its Metabolites Impact Immune Responses in COVID-19 and Its Complications. Gastroenterology. 2023 Feb;164(2):272-288. doi: 10.1053/j.gastro.2022.09.024. Epub 2022 Sep 23. PMID 36155191
- [Background] Sherif ZA, Gomez CR, Connors TJ, Henrich TJ, Reeves WB; RECOVER Mechanistic Pathway Task Force. Pathogenic mechanisms of post-acute sequelae of SARS-CoV-2 infection (PASC). Elife. 2023 Mar 22;12:e86002. doi: 10.7554/eLife.86002. PMID 36947108
- [Background] Sukocheva OA, Maksoud R, Beeraka NM, Madhunapantula SV, Sinelnikov M, Nikolenko VN, Neganova ME, Klochkov SG, Amjad Kamal M, Staines DR, Marshall-Gradisnik S. Analysis of post COVID-19 condition and its overlap with myalgic encephalomyelitis/chronic fatigue syndrome. J Adv Res. 2022 Sep;40:179-196. doi: 10.1016/j.jare.2021.11.013. Epub 2021 Nov 26. PMID 36100326
- [Background] Xu E, Xie Y, Al-Aly Z. Long-term gastrointestinal outcomes of COVID-19. Nat Commun. 2023 Mar 7;14(1):983. doi: 10.1038/s41467-023-36223-7. PMID 36882400
- [Background] Zuo T, Zhang F, Lui GCY, Yeoh YK, Li AYL, Zhan H, Wan Y, Chung ACK, Cheung CP, Chen N, Lai CKC, Chen Z, Tso EYK, Fung KSC, Chan V, Ling L, Joynt G, Hui DSC, Chan FKL, Chan PKS, Ng SC. Alterations in Gut Microbiota of Patients With COVID-19 During Time of Hospitalization. Gastroenterology. 2020 Sep;159(3):944-955.e8. doi: 10.1053/j.gastro.2020.05.048. Epub 2020 May 20. PMID 32442562

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT05874089/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT05874089/ICF_001.pdf